CLINICAL TRIAL: NCT00851370
Title: Exploratory Study of Xolair (Omalizumab)to Improve Outcomes in Patients With COPD and Elevated IgE Levels, and Positive RAST or Skin Prick Tests
Brief Title: Exploratory Study of Xolair in Chronic Obstructive Pulmonary Disease in Patients With Elevated IgE Levels
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to find eligible subjects- study closed
Sponsor: National Jewish Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NJ-241
Record Dates: First submitted 2009-02-04; First posted 2009-02-25 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omalizumab (Experimental)
  Interventions: Drug: Omalizumab (Xolair)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab (Xolair) — Bi-weekly
  Other Names: Xolair
  Arms: Omalizumab
Drug: Placebo — Bi-Weekly
  Arms: Placebo

SUMMARY:
The objective is to conduct an exploratory study on the effect of Omalizumab on COPD patients with elevated IgE. Exploratory outcomes include to determine whether Omalizumab use: reduces exacerbations in COPD patients; or improves rescue medication use, decreases ICS use, modified Medical Research Council (MMRC) dyspnea score, St. George's Respiratory Questionnaire (SGRQ), 6-minute walk distance (6MWD), forced expiratory volume at one second (FEV1)(the latter 3 with BMI make up the BODE score), residual volume (RV), total lung capacity (TLC), exhaled nitric oxide (ENO), and determination C-reactive protein (CRP).

ELIGIBILITY:
Inclusion Criteria:

* Smoking-related COPD and aged between 40 and 70 yrs.
* Total IgE of 30-700 IU and a positive RAST or skin prick test result to one or more perennial environmental allergens (e.g. dust mite (Dermatophagoides farinae, Dermatophagoides pteronyssinus), cockroach, dog, or cat.)
* Any race or sex; women with childbearing potential are required to use an acceptable method for birth control and have a negative pregnancy test
* History of ≥2 exacerbations during 2 yrs previous to the enrollment date
* An exacerbation will be defined as an increase or new onset of more than one of the following: cough, sputum, wheezing, dyspnea, or chest tightness with a duration of at least 3 days requiring antibiotic or systemic steroid treatment. The severity of an exacerbation will be determined by the following:
* Mild: Home management, with or without contacting a health care provider, or unscheduled office visit
* Moderate: Requiring a visit to an emergency department
* Severe: Requiring hospitalization
* Very Severe: Requiring intubation and medical ventilation
* Post-bronchodilator FEV1 30-64% of predicted; the first 5 subjects enrolled will be required to have post-bronchodilator FEV1 50-64%
* Post-bronchodilator FEV1/FVC < 0.7
* Smokers or ex-smokers with at least a 20 pack-year smoking history
* Able to communicate meaningfully with the study personnel and to understand and read fluently in English
* Written informed consent;
* BODE score 3-10.

Exclusion Criteria:

* History of Omalizumab use
* Evidence of illicit drug use or abuse of alcohol.
* Women of childbearing potential not using the contraception method(s) specified in this study (specify), as well as women who are breastfeeding
* Known sensitivity to study drug(s) or class of study drug(s)
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (specify as required)
* Use of any other investigational agent in the last 30 days
* Continuous treatment with oral corticosteroids
* Participating in another trial within 3 months prior to the beginning of the study
* Non-compliance in taking medications
* Planned for lung transplantation at the time of admission to the study or expected to be transplanted within 3 yrs
* Alpha-1-antitrypsin deficiency
* Cystic fibrosis
* Bronchiectasis
* History of infection or active infection due to Mycobacterium tuberculosis
* Pneumoconiosis
* Pulmonary restriction due to any other pulmonary disease, apart from the one concerned with the study population
* Congestive heart failure class 2 or more of the New York Heart Association (NYHA)
* Reduced life expectancy due to other disease (defined as having an expected mortality of ≥25% five years from enrollment)
* Current use of ß-blockers

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
COPD Exacerbations | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Russell P Bowler, MD, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Cazzola M, Dahl R. Inhaled combination therapy with long-acting beta 2-agonists and corticosteroids in stable COPD. Chest. 2004 Jul;126(1):220-37. doi: 10.1378/chest.126.1.220. PMID 15249466
- [Background] Bonay M, Bancal C, Crestani B. The risk/benefit of inhaled corticosteroids in chronic obstructive pulmonary disease. Expert Opin Drug Saf. 2005 Mar;4(2):251-71. doi: 10.1517/14740338.4.2.251. PMID 15794718
- [Background] Imfeld S, Bloch KE, Weder W, Russi EW. The BODE index after lung volume reduction surgery correlates with survival. Chest. 2006 Apr;129(4):873-8. doi: 10.1378/chest.129.4.873. PMID 16608932